CLINICAL TRIAL: NCT07157345
Title: A Study on the Safety, Tolerability, and Efficacy of PDR-001 Injection for Bilateral Stereotactic Subthalamic Nucleus (STN) Clearance of α-synuclein
Brief Title: Testing if PDR-001 Can Safely and Effectively Remove Harmful Brain Protein in Parkinson's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V1.0/2025-07-06
Record Dates: First submitted 2025-08-05; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease (PD)
Keywords: PDR-001; Parkinson disease
MeSH Terms: conditions — Parkinson Disease | interventions — spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- primary parkinson's disease (Experimental): PDR-001 injection, inject once, 0.4 milliliters each time
  Interventions: Drug: PDR001

INTERVENTIONS:
Drug: PDR001 — This drug was packaged into AAV9 capsids and delivered via bilateral stereotaxic injection into the subthalamic nucleus

SUMMARY:
Parkinson's disease (PD) poses a severe threat to human health, and its incidence is rising year by year. Current therapeutic options are limited by significant shortcomings. Pathological aggregation of α-synuclein and the consequent death of dopaminergic neurons are the primary drivers of PD pathogenesis. While siRNA-mediated knockdown of α-synuclein can offer some protection to dopaminergic neurons, its clinical utility is hampered by low cellular uptake, off-target effects, and transient activity. These drawbacks underscore the urgent need for novel strategies that can efficiently and specifically degrade α-synuclein to delay or even halt PD progression.

Our prior work identified tat-βsyn-deg (PDR-001), a three-segment peptide that selectively targets α-synuclein. When packaged into AAV9 capsids and delivered via bilateral stereotaxic injection into the subthalamic nucleus, this peptide effectively reduces α-synuclein within the target region. Pre-clinical studies in both human-α-synuclein-expressing mice and non-human primate models of PD have demonstrated robust α-synuclein clearance and marked improvements in motor deficits (see Research Foundation).

The present project will advance PDR-001 into first-in-human studies to evaluate safety and explore preliminary efficacy. Unlike conventional symptomatic therapies, this approach targets the root cause of PD, setting the stage for disease-modifying treatment. Successful translation would establish a new therapeutic paradigm capable of slowing or preventing PD progression.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion in this clinical study, all of the following criteria must be met:

1. Clinically confirmed diagnosis of primary PD (in accordance with the 2016 Chinese Diagnostic Criteria for Parkinson's Disease or the 2015 MDS Clinical Diagnostic Criteria for primary PD);
2. Age 40-65 years (inclusive) at screening, either sex;
3. Disease duration ≤ 5 years;
4. Hoehn & Yahr stage ≤ 2 in the "off" state.

Exclusion Criteria:

Exclusion Criteria

1. Atypical or secondary parkinsonian syndromes (e.g., Parkinson-plus syndromes, hereditary parkinsonism, drug-induced parkinsonism, etc.).
2. Contra-indications to surgery, or any prior intracranial procedure such as deep-brain stimulation, pallidotomy, or other extrapyramidal surgery, or any other neurosurgical intervention deemed by the investigator to interfere with study participation.
3. Previous neuroimaging revealing structural brain abnormalities, cerebral vascular malformations, intracranial tumors, risk of intracranial hemorrhage, traumatic brain injury, or other significant findings.
4. Mini-Mental State Examination (MMSE) score < 24.
5. Patient Health Questionnaire-9 (PHQ-9) score ≥ 16.
6. Abnormal hepatic or renal function: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 × upper limit of normal (ULN), or serum creatinine (Cr) > 1.5 × ULN.
7. Coagulation disorders or current use of anticoagulants.
8. Positive screening for infectious diseases:

   * Hepatitis B surface antigen (HBsAg) or Hepatitis B virus DNA (HBV-DNA) positive;
   * Hepatitis C virus RNA (HCV-RNA) positive;
   * Human immunodeficiency virus (HIV) positive;
   * Positive syphilis serology.
9. Currently receiving antiviral therapy for hepatitis B or C.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
PDR-001 treatment-related adverse events as assessed by CTCAE v5.0 | From enrollment to the end of treatment at 52 weeks
  CTCAE 5.0 records the severity of adverse events, which is divided into grades 1 to 5
Titer levels of capsid neutralizing antibodies and binding antibodies against recombinant adeno-associated virus (rAAV) in serum | From enrollment to the end of treatment at 52 weeks
  Record the titer changes before and after treatment
Titer of rAAV vectors in whole blood | From enrollment to the end of treatment at 52 weeks
  Record the titer changes before and after treatment

SECONDARY OUTCOMES:
Evaluation of the use of antiparkinsonian drugs will be assessed using the Levodopa Equivalent Daily Dose (LEDD) | From enrollment to the end of treatment at 52 weeks
  The total daily dose of antiparkinsonian medication (converted to LEDD, mg/day) will be calculated and compared before and after treatment. A decrease in LEDD indicates reduced drug burden (better outcome), while an increase indicates greater drug requirement (worse outcome).
Treatment efficacy will be evaluated using the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | From enrollment to the end of treatment at 52 weeks
  This scale has a total score range of 0 to 260, with higher scores indicating more severe motor and non-motor symptoms (worse outcome). Changes in scores before and after treatment will be recorded.
Treatment efficacy will be evaluated using the Patient Global Impression - Improvement scale (PGI-I) | From enrollment to the end of treatment at 52 weeks
  This is a 7-point scale ranging from 1 ("very much improved") to 7 ("very much worse"), with lower scores indicating greater improvement (better outcome). Changes in scores before and after treatment will be recorded.
Treatment efficacy will be evaluated using the Clinical Global Impression - Improvement scale (CGI-I) | From enrollment to the end of treatment at 52 weeks
  This is a 7-point scale ranging from 1 ("very much improved") to 7 ("very much worse"), with lower scores indicating greater clinical improvement (better outcome). Changes in scores before and after treatment will be recorded.
Treatment efficacy will be evaluated using the Mini-Mental State Examination (MMSE) | From enrollment to the end of treatment at 52 weeks
  The total score ranges from 0 to 30, with higher scores indicating better cognitive function (better outcome). Changes in scores before and after treatment will be recorded.
Treatment efficacy will be evaluated using the Hamilton Depression Rating Scale (HAM-D, 17-item version) | From enrollment to the end of treatment at 52 weeks
  The total score ranges from 0 to 52, with higher scores indicating more severe depressive symptoms (worse outcome). Changes in scores before and after treatment will be recorded.
Change in anxiety symptoms as measured by the Hamilton Anxiety Rating Scale (HAM-A) | From enrollment to the end of treatment at 52 weeks
  The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered scale with scores ranging from 0 to 56, where higher scores indicate greater severity of anxiety symptoms. Treatment efficacy will be evaluated by the change in HAM-A total score from baseline to 52 weeks
Change in sleep-related problems as measured by the Parkinson's Disease Sleep Scale-2 (PDSS-2) | From enrollment to the end of treatment at 52 weeks
  PDSS-2 is a 15-item questionnaire. The total score ranges from 0 to 60, with higher scores indicating worse sleep-related problems. Treatment efficacy will be evaluated by the changes in PDSS-2 from baseline to 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT07157345/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT07157345/ICF_001.pdf